CLINICAL TRIAL: NCT04677517
Title: Impact of Microphone Positioning on Auditory Performance in Cochlear Implant Users
Acronym: MICLO
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The project has been replaced by anotherone with a different regulatory qualification
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 69HCL20_1013
Record Dates: First submitted 2020-12-16; First posted 2020-12-21 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Cochlear Prosthesis Implantation
Keywords: Cochlear implants users; microphone; virtual reality; spatial hearing perception

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Implanted patients (Experimental): All the participants are patients with post-lingual deafness and fitted with cochlear implants
  Interventions: Device: Modification of active microphone positioning; Behavioral: SPHERE protocol; Behavioral: French Matrix Test; Behavioral: Quality of life questionnaire; Behavioral: Likert scale

INTERVENTIONS:
Device: Modification of active microphone positioning — Patient will pass the experimental tests described above with 3 different active microphone positions :
  * on the cochlear implant processor;
  * on the antenna
  * in front of the external ear canal
  Patient will pass the tests 1 week after each microphone position change, so that they can get used to the new position in their everyday life.
Behavioral: SPHERE protocol — Patient's 3D localization in noise will be assessed thnks to a 3D localization system called SPHERE based on virtual reality.
  Data from spatial hearing perception will be recorded in three-dimensional space (azimuth, elevation, and depth). First, the pointing error will be computed separately for azimuth, elevation, and depth, in terms of constant error (absolute and signed) and variable error. Then, these separate errors will be combined into a cumulative error "3d-D" (the 3d-D value), hence summarizing all three space dimensions, and taking into account absolute and variable error in one measure.
Behavioral: French Matrix Test — This test assesses the intelligibility threshold defined as the noise level (in decibels) for which the subject can repeat 50% of the words heard (in dichotic listening), resulting in an Speech Recognition Threshold (SRT) value
Behavioral: Quality of life questionnaire — The Speech, Spatial and Qualities of Hearing Scale short-form with 15 items (SSQ15) questionnaire is performed in order to evaluate auditory abilities of patients in different daily life situations.
Behavioral: Likert scale — This subjective evaluation will be added to evaluate difficulties and self-confidence felt by participants during the SPHERE protocol and the French Matrix Test.

SUMMARY:
The construction of our auditory space requires several prerequisites, including localization abilities in 3D (azimuth, elevation and distance). These abilities rely on the proper development and functionality of the auditory system to extract various acoustic cues from our environment. Extraction and analysis of these auditory cues are based on the synchronous use of ears, called binaurality. Other natural behaviours are useful to precisely determine the location of a sound source: visual information and head movements.

The slightest anatomical-functional change (e.g. unilateral hearing loss, malformation of the pinna) can disturb spatial hearing abilities. Many patients with hearing loss are fitted with a hearing aid (HA) or a cochlear implant (CI) to ensure the best speech understanding. However, this auditory rehabilitation remains insufficient to restore a good perception of spatial hearing. One of the key point to improve sound localization seems to be microphone positioning on hearing aids. Several questions remain on the optimal microphone positioning.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 75 inclusive
* Regular follow-up in the Ear Nose and Throat department of the Edouard Herriot hospital in Lyon
* Post-lingual deafness
* Fitted with two Advanced Bionics (AB) cochlear implants (Naïda Q70 or Naïda Q90 processor) Or fitted with one AB cochlear implant and a contralateral hearing aid
* Fitted with the latest implant for more than 1 year
* Normal or corrected vision
* Able to understand experimental instructions
* Affiliated with a social security scheme

Exclusion Criteria:

* Oculomotor disorder
* Bilateral vestibular areflexia
* Adult subject to a legal protection measure (guardianship, curatorship)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-12-01 (Estimated); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in 3d-D value at day 7 | Baseline and day 7
  We will compare 3d-D values obtained with baseline microphone position (at day 0) and 1 week after the first microphone positioning change. Baseline microphone position is defined as the usual position at inclusion and might vary from one patient to another. Combined with change in SRT values and SSQ15 scores, these results will allow us to assess the effect of microphones positioning on spatial auditory performance.
Change from baseline in 3d-D value at day 14 | Baseline and day 14
  We will compare 3d-D values obtained with baseline microphone position (at day 0) and 1 week after the second microphone positioning change. Baseline microphone position is defined as the usual position at inclusion and might vary from one patient to another. Combined with change in SRT values and SSQ15 scores, these results will allow us to assess the effect of microphones positioning on spatial auditory performance.
Change from baseline in SRT value at day 7 | Baseline and day 7
  We will compare SRT values obtained with baseline microphone position (at day 0) and 1 week after the first microphone positioning change. Baseline microphone position is defined as the usual position at inclusion and might vary from one patient to another. Combined with change in 3d-D values and SSQ15 scores, these results will allow us to assess the effect of microphones positioning on spatial auditory performance.
Change from baseline in SRT value at day 14 | Baseline and day 14
  We will compare SRT values obtained with baseline microphone position (at day 0) and 1 week after the second microphone positioning change. Baseline microphone position is defined as the usual position at inclusion and might vary from one patient to another. Combined with change in 3d-D values and SSQ15 scores, these results will allow us to assess the effect of microphones positioning on spatial auditory performance.
Change from baseline in SSQ15 score at day 7 | Baseline and day 7
  We will compare SSQ15 scores obtained with baseline microphone position (at day 0) and 1 week after the first microphone positioning change. Baseline microphone position is defined as the usual position at inclusion and might vary from one patient to another. Combined with change in 3d-D values and SRT values, these results will allow us to assess the effect of microphones positioning on spatial auditory performance.
Change from baseline in SSQ15 score at day 14 | Baseline and day 14
  We will compare SSQ15 scores obtained with baseline microphone position (at day 0) and 1 week after the second microphone positioning change. Baseline microphone position is defined as the usual position at inclusion and might vary from one patient to another. Combined with change in 3d-D values and SRT values, these results will allow us to assess the effect of microphones positioning on spatial auditory performance.

CONTACTS AND LOCATIONS:
Overall Officials: Eric TRUY, Professor, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Hôpital Edouard Herriot - service ORL, Lyon, France